CLINICAL TRIAL: NCT07364981
Title: Gaze Contingent Attentional Reinforcement Treatment of MDD
Brief Title: Gaze Contingent Attentional Reinforcement in Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Amit Lazarov, Professor of Psychology, School of Psychological Sciences, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAU-MDD
Record Dates: First submitted 2025-12-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD; attention allocation; positive reinforcement; negative reinforcement
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaze contingent negative reinforcement (Active Comparator): participants will receive gaze-contingent negative reinforcement according to their viewing patterns
  Interventions: Behavioral: Aversive white noise
- Gaze contingent positive reinforcement (Placebo Comparator): participants will receive gaze-contingent positive reinforcement according to their viewing patterns
  Interventions: Behavioral: Music reward

INTERVENTIONS:
Behavioral: Aversive white noise — Participants will receveve gaze-contingent negative-reinforcement feedback according to their viewing patterns, such that when gazing at the target stimuli (i.e., happy faces) the noise will stop.
  Arms: Gaze contingent negative reinforcement
Behavioral: Music reward — Participants will receive gaze-contingent music-reward according to their viewing patterns, such that when gazing at the target stimuli (i.e., happy faces) the music will play.
  Arms: Gaze contingent positive reinforcement

SUMMARY:
The main objective of this randomized controlled trial is to evaluate whether a gaze-contingent feedback task using negative reinforcement can serve as an effective attention-modification procedure and contribute to the treatment of Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This randomized controlled trial uses a gaze-contingent attentional reinforcement task to modify attention allocation patterns to emotional stimuli in participants with Major Depressive Disorder. Specifically, participants will undergo 4 training sessions, during which either negative reinforcement (aversive white noise will be heard when gazing at sad faces) or positive reinforcement (music will be heard when gazing at happy faces) will be used to divert participants' gaze toward happy faces and away from sad faces. Depressive symptoms severity will be assessed before and after training (post-training and 3-month follow up) to examine changes (reduction) in symptom severity from before to after the intervention. Attention allocation will be assessed during training (i.e. online learning) as well as before and after training (i.e. transfer of learning).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of MDD
* MADRS>=7
* Normal or corrected-t-normal vision

Exclusion Criteria:

* Present or past psychosis, manic or hypomanic episode, PTSD
* High suicidal ideation or behavior
* Severe alcohol or cannabis use disorder, and/or any severity of other substance use disorder (exepct nicotine use)
* Pharmacological treatment if not stabilized for at least three months or concurrent psychotherapy
* Current unstable or untreated medical illness
* Current or past organic mental disorder, seizure or brain injury
* Eye-tracking calibration difficulties
* Post-ECT treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
MADRS- diagnostic interview scores | Post-treatment (1 week after treatment completion) and 3-month follow up
  Change from baseline- the Montgomery Asberg Depression Rating scale is a clinician-administered scale that includes 10 items that measure the severity of depressive symptoms. Each of the 10 items is scored on a 7-point scale (0-6). The total score, ranging from 0 to 60 is used to assess severity.

SECONDARY OUTCOMES:
PHQ-9 - self report measure | Post-treatment (1 week after treatment completion) and 3-month follow up
  Change from baseline- the Patient Health Questionnaire-9 is a nine-question self-report questionnaire to assess the severity of depression based on symptoms over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day). The overal score ranges from 0-27, indicating depression severity.

OTHER OUTCOMES:
Attention Allocation | Post-treatment (1 week after treatment completion) and 3-month follow up
  Changes from baseline- attention allocation towards the target stimuli (happy faces) compared to the non-target stimuli (sad faces).
M.I.N.I diagnosis- diagnostic interview | Post-treatment (1 week after treatment completion) and 3-month follow up
  Changes in the Mini-International Neuropsychiatric Interview diagnosis. The M.I.N.I. is a structured diagnostic interview for DSM-5 and ICD-11 psychiatric disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Lazarov, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No